CLINICAL TRIAL: NCT00006050
Title: Chemotherapy Intra-Arterial Hepatic With Oxaliplatin Combined With Leucovorin Calcium and Fluorouracil IV
Brief Title: Combination Chemotherapy in Treating Patients With Colorectal Cancer That Has Spread to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068072; FRE-FNCLCC-98012-PAC-ACCORD-04; EU-20017
Record Dates: First submitted 2000-07-05; First posted 2004-02-02 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: isolated perfusion
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of liver perfusion using oxaliplatin plus leucovorin and fluorouracil given by infusion in treating patients who have colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and tolerance of oxaliplatin by hepatic perfusion combined with intravenous leucovorin calcium and fluorouracil in patients with liver metastases from colorectal cancer.

OUTLINE: Patients receive oxaliplatin by hepatic perfusion over 2 hours on day 1 plus leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity. If a good response is achieved after 8 courses of chemotherapy, patients may undergo surgical resection of metastases.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven colorectal cancer metastatic to the liver Unresectable disease Less than 50% invasion of the liver Measurable disease No prior irradiation Largest diameter at least 20 mm No detectable extrahepatic disease

PATIENT CHARACTERISTICS: Age: Under 75 Performance status: WHO 0-2 Life expectancy: Greater than 2 months Hematopoietic: WBC at least 4,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 35 micromoles/L Renal: Creatinine less than 130 micromoles/L Cardiovascular: No severe cardiac insufficiency Pulmonary: No respiratory disease that would preclude study Other: No other serious illness that would preclude study No psychological illness that would preclude study No peripheral neuropathy No prior malignancy not considered cured Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior intravenous oxaliplatin No more than 1 prior regimen of intravenous chemotherapy for metastatic disease Primary chemotherapy of fluorouracil allowed if stable or progressive disease No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04-04 (Actual); Primary Completion 2001-12-31 (Actual); Study Completion 2003-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Ducreux M, Ychou M, Laplanche A, Gamelin E, Lasser P, Husseini F, Quenet F, Viret F, Jacob JH, Boige V, Elias D, Delperro JR, Luboinski M; gastrointestinal group of the Federation Nationale des Centres de Lutte Contre le Cancer. Hepatic arterial oxaliplatin infusion plus intravenous chemotherapy in colorectal cancer with inoperable hepatic metastases: a trial of the gastrointestinal group of the Federation Nationale des Centres de Lutte Contre le Cancer. J Clin Oncol. 2005 Aug 1;23(22):4881-7. doi: 10.1200/JCO.2005.05.120. Epub 2005 Jul 11. PMID 16009952